CLINICAL TRIAL: NCT00394862
Title: Efficacy of Weekly Versus Daily Folic Acid Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Reynaldo Martorell, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 205-2004
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Neural Tube Defects
MeSH Terms: conditions — Neural Tube Defects | interventions — Geritol

INTERVENTIONS:
Drug: multivitamin

SUMMARY:
Investigate the efficacy of weekly versus daily of folic acid supplementation on improving folate, vitamin B12,

DETAILED DESCRIPTION:
460 women of a rural community in the western highlands of Guatemala were recruited for participation in the double-blinded study led by Emory University and the Institute of Nutrition of Central America and Panama (INCAP). The women were randomly assigned one of 4 vitamin treatments containing different levels of folic acid, Vitamin B12, iron and zinc. The treatments were as follows:

1. weekly dose of folic acid at 5000ug, iron at 120 mg, zinc at 30mg, and B12 at 16.8 ug;
2. weekly dose of folic acid at 2800ug, iron at 120mg, zinc at 0mg and B12 at 16.8ug;
3. daily dose of folic acid at 400ug, iron at 60mg, zinc at 15mg, B12 at 2.4ug; and
4. daily dose of folic acid at 200ug, iron at 50mg, zinc at 0mg, and B12 at 2.4ug.

The women, aged 15-49, received the vitamins daily for 3 months. Anthropometric data and blood samples were taken at baseline and post-supplementation. The participants also completed a series of dietary interviews at baseline and post-intervention. No pregnant or lactating mothers were admitted into the study, nor severely anemic females. Blood samples were sent to the National Laboratory in Cuernavaca, Mexico, for analysis of serum folate levels.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged 15-49

Exclusion Criteria:

* pregnant
* lactating less than 3 months
* severely anemic

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 460
Dates: Start 2006-01; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
serum folate level
red blood cell folate

SECONDARY OUTCOMES:
homocysteine
ferritin
serum zinc
serum B12
blood pressure
depression

CONTACTS AND LOCATIONS:
Overall Officials: Reynaldo Martorell, PHD, MPH, Principal Investigator — Emory University